CLINICAL TRIAL: NCT05813717
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single Doses of BMS-986325 in Healthy Japanese Participants
Brief Title: A Study to Evaluate the Safety, Tolerability, Drug Levels, and Drug Effects of BMS-986325 in Healthy Japanese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IM039-1001
Record Dates: First submitted 2023-04-03; First posted 2023-04-14 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-10

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort J1 (Experimental)
  Interventions: Drug: BMS-986325; Drug: Placebo
- Cohort J2 (Experimental)
  Interventions: Drug: BMS-986325; Drug: Placebo
- Cohort J3 (Experimental)
  Interventions: Drug: BMS-986325; Drug: Placebo

INTERVENTIONS:
Drug: BMS-986325 — Specified dose on specified days
Drug: Placebo — Specified dose on specified days

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of BMS-986325 in healthy Japanese participants

ELIGIBILITY:
Inclusion Criteria:

* Participants must be ethnically Japanese (both biological parents are ethnically Japanese).
* Healthy male and female participants as determined by no clinically significant deviation from normal in medical history, physical examination, 12-lead ECGs, or clinical laboratory determinations.
* Body mass index (BMI) between 18 and 30 kg/m2, inclusive, at screening.

Exclusion Criteria:

* Any significant acute or chronic medical illness.
* Any major surgery within 4 weeks prior to study drug administration, or any surgery planned during the course of the study.
* Any history of known or suspected congenital or acquired immunodeficiency state or condition that would compromise the participant's immune status (eg, history of splenectomy).

Other protocol-defined inclusion/exclusion criteria apply.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2023-04-10 (Actual); Primary Completion 2023-10-02 (Actual); Study Completion 2023-10-02 (Actual)

PRIMARY OUTCOMES:
Number of participants with Adverse events | Up to day 92
Number of participants with clinical laboratory abnormalities | Up to day 64
Number of participants with vital sign abnormalities | Up to day 64
Number of participants with ECG abnormalities | Up to day 64
Number of participants with physical examination abnormalities | Up to day 64

SECONDARY OUTCOMES:
Serum concentrations of BMS-986325 | Up to day 64
Maximum observed serum concentration (Cmax) | Up to day 64
Time of maximum observed serum concentration (Tmax) | Up to day 64
Area under the serum concentration-time curve from time zero to time of last quantifiable concentration (AUC(0-T)) | Up to day 64
Pharmacokinetics/pharmacodynamic (receptor occupancy) (PK/PD (RO)) correlation | Up to day 64
  Receptor occupancy assays are measured by BMS-986325 binding with fluorescently conjugated antibodies on B cells. Receptor occupancy is calculated as a ratio of fluorescence intensity using unchallenged samples over fluorescence intensity using saturated samples.
Absolute Bioavailability (F) of BMS-986325 | Up to day 64
  Measured as a percentage
Number of Participants With Anti-Drug Antibody Response | Up to day 64

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution - 0001, Cypress, California, United States

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm